CLINICAL TRIAL: NCT00706992
Title: Transfer of Autologous T Cells Transduced With the Anti-MART-1 F5 T Cell Receptor in High Risk Melanoma
Brief Title: Anti-MART-1 F5 Lymphocytes to Treat High-Risk Melanoma Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: <11 subjects were enrolled to each Arm
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Steven Rosenberg, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 080162; 08-C-0162
Record Dates: First submitted 2008-06-27; First posted 2008-06-30 (Estimated); Results first posted 2013-03-19 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Melanoma
Keywords: MART-1 Peptide; Melanoma; Adjuvant Therapy; Gene Therapy; T Cell Persistence
MeSH Terms: conditions — Melanoma | interventions — Protein Subunit Vaccines; aldesleukin; incomplete Freund's adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Arm I - Adj-4 A2 F5 cells (Experimental): Patients receive anti-MART-1 F5 TCR-transduced peripheral blood lymphocytes (PBLs) intravenously (IV) over 20-30 minutes on day 0. 1 x 10e9 to 5 x 10e10 IV.
  Interventions: Biological: autologous anti-MART-1 F5 T-cell receptor gene-engineered peripheral blood lymphocytes
- Arm II-Adj-4 A2 F5 cells + MART-1:26-35(27L) Peptide (Experimental): Patients receive anti-MART-1 F5 TCR-transduced PBLs as in arm I and MART-1:26-35(27L) peptide vaccine emulsified in Montanide ISA-51 subcutaneously (SC) on days 0 and 30. 1 x 10e9 to 5 x 10e10 IV + 1.0 mg peptide subcutaneously.
  Interventions: Biological: MART-1:26-35(27L) peptide vaccine; Biological: autologous anti-MART-1 F5 T-cell receptor gene-engineered peripheral blood lymphocytes; Biological: incomplete Freund's adjuvant
- Arm III-Adj-4 A2 F5 cells + SQ IL-2 (Experimental): Patients receive anti-MART-1 F5 TCR-transduced PBLs as in arm I and aldesleukin SC on days 0-4. 1 x 10e9 to 5 x 10e10 IV + IL-2 (based on body weight) 125,000 IU/kg/day subcutaneously.
  Interventions: Biological: Aldesleukin; Biological: autologous anti-MART-1 F5 T-cell receptor gene-engineered peripheral blood lymphocytes
- Arm IV-Adj-4 A2 F5 cells + MART-1:26-35(27L) Peptide+SQ IL-2 (Experimental): Patients receive anti-MART-1 F5 TCR-transduced PBLs as in arm I, MART-1:26-35(27L) peptide vaccine emulsified in Montanide ISA-51 as in arm II, and aldesleukin as in arm III. 1 x 10e9 to 5 x 10e10 IV + 1.0 mg peptide subcutaneously + IL-2 (based on body weight) 125,000 IU/kg/day subcutaneously.
  Interventions: Biological: MART-1:26-35(27L) peptide vaccine; Biological: Aldesleukin; Biological: autologous anti-MART-1 F5 T-cell receptor gene-engineered peripheral blood lymphocytes; Biological: incomplete Freund's adjuvant
- Arm V-Adj-4 A2 F5 cells + ALVAC MART-1:26-35(27L) Vaccine (Experimental): Patients receive anti-MART-1 F5 TCR-transduced PBLs IV over 20-30 minutes on day 0, and ALVAC-MART-1 vaccine SC on days 0 and 14. 1 x 10e9 to 5 x 10e10 IV + ALVAC vaccine 0.5 ml containing target dose of 10e7 CCID50 (with a range of approximately 10^6.4 to 10^7.9/mL subcutaneously (total of 4 x 10e7 CCID50/2 mL).
  Interventions: Biological: ALVAC-MART-1 vaccine; Biological: autologous anti-MART-1 F5 T-cell receptor gene-engineered peripheral blood lymphocytes
- Arm VI-Adj-4 A2 F5 cells + ALVAC MART-1 VAccine + SQ IL-2 (Experimental): Patients receive anti-MART-1 F5 TCR-transduced PBLs and ALVAC-MART-1 vaccine as in arm V, and low-dose aldesleukin SC on days 0-4. 1 x 10e9 to 5 x 10e10 IV + ALVAC vaccine 0.5 ml containing target dose of 10e7 CCID50 (with a range of approximately 10^6.4 to 10^7.9/mL subcutaneously (total of 4 x 10e7 CCID50/2 mL)+ 125,000 IU/kg/day subcutaneously.
  Interventions: Biological: ALVAC-MART-1 vaccine; Biological: autologous anti-MART-1 F5 T-cell receptor gene-engineered peripheral blood lymphocytes
- Arm VII-Adj-4 A2 ALVAC MART-1:26-35(27L) Vaccine (Experimental): Patients receive ALVAC-MART-1 vaccine SC on days 0 and 14. ALVAC vaccine 0.5 ml containing target dose of 10e7 CCID50 (with a range of approximately 10^6.4 to 10^7.9/mL subcutaneously (total of 4 x 10e7 CCID50/2 mL).
  Interventions: Biological: ALVAC-MART-1 vaccine; Biological: Aldesleukin; Biological: autologous anti-MART-1 F5 T-cell receptor gene-engineered peripheral blood lymphocytes

INTERVENTIONS:
Biological: ALVAC-MART-1 vaccine — Given subcutaneously
  Arms: Arm V-Adj-4 A2 F5 cells + ALVAC MART-1:26-35(27L) Vaccine; Arm VI-Adj-4 A2 F5 cells + ALVAC MART-1 VAccine + SQ IL-2; Arm VII-Adj-4 A2 ALVAC MART-1:26-35(27L) Vaccine
Biological: MART-1:26-35(27L) peptide vaccine — Given subcutaneously
  Arms: Arm II-Adj-4 A2 F5 cells + MART-1:26-35(27L) Peptide; Arm IV-Adj-4 A2 F5 cells + MART-1:26-35(27L) Peptide+SQ IL-2
Biological: Aldesleukin — Given subcutaneously
  Arms: Arm III-Adj-4 A2 F5 cells + SQ IL-2; Arm IV-Adj-4 A2 F5 cells + MART-1:26-35(27L) Peptide+SQ IL-2; Arm VII-Adj-4 A2 ALVAC MART-1:26-35(27L) Vaccine
Biological: autologous anti-MART-1 F5 T-cell receptor gene-engineered peripheral blood lymphocytes — Given intravenously (IV)
Biological: incomplete Freund's adjuvant — Given subcutaneously
  Arms: Arm II-Adj-4 A2 F5 cells + MART-1:26-35(27L) Peptide; Arm IV-Adj-4 A2 F5 cells + MART-1:26-35(27L) Peptide+SQ IL-2

SUMMARY:
Background:

* Melanoma antigen recognized by T cells (MART-1) is a gene that is present in melanoma cells.
* This study tests an experimental treatment that uses the patient's own lymphocytes (type of white blood cell), which are specially selected and genetically modified with a gene called anti-MART-1 transduced cells (F5) to target and destroy their tumor. Some of the cells are given as an infusion and others are given as a vaccine.
* The anti-MART-1 F5 cells are currently being studied in other patients in combination with chemotherapy and IL-2 (aldesleukin) therapy.

Objectives:

-To determine if the anti-MART-1 F5 treatment can improve the immune system's ability to shrink tumors and to prevent melanoma from recurring.

Eligibility:

* Patients 18 years of age and older whose melanoma has been removed and are currently disease-free, but who are at risk for recurrence.
* Patients who do not have ocular or mucosal melanoma.
* Patients with tissue type human leukocyte antigens (HLA-A)*0201).

Design:

* Workup: Patients have scans, x-rays, laboratory tests, other tests as needed and leukapheresis, a procedure for collecting white cells to modify in the laboratory and later reinfuse into the patient.
* Patients are assigned to one of four study groups:

  * Group 1 receives anti-MART-1 F5 cells by 30-minute infusion through a vein on day 0.
  * Group 2 receives anti-MART-1 F5 cells on day 0 followed by injections of MART-1 vaccine, which contains MART-1 and an oil-based liquid called Montanide ISA-51 VG. The vaccine is repeated on day 30.
  * Group 3 receives anti-MART-1 F5 cells on day 0 followed by injections of low-dose IL-2 for 5 days (days 0-4).
  * Group 4 receives anti-MART-1 F5 cells on day 0 followed by MART-1 vaccine and low-dose IL-2 for 5 days. The vaccine is repeated on day 30.
* Recovery: Patients are monitored closely and given medicines to prevent or treat any side effects of therapy.
* Leukapheresis: Patients undergo leukapheresis at 1 and 3 months after therapy to collect cells to examine the effects of the treatment on the immune system.
* Follow-up: Patients return to National Institutes of Health (NIH) 35 days after completing treatment and then at 3 months and every 6 months thereafter for evaluation with a physical examination, review of side effects, laboratory tests and scans. They have blood tests at 3, 6 and 12 months after treatment and then once a year after that. A biopsy may be requested after treatment ends to examine the effects of treatment on the immune system. All patients return to NIH for a physical examination once a year for 5 years and then complete a follow-up questionnaire for another 10 years.

DETAILED DESCRIPTION:
Background:

We have engineered human peripheral blood lymphocytes (PBLs) to express an anti-MART-1 T-cell receptor (TCR) that recognizes an HLA-A*0201 restricted epitope derived from the tumor infiltrating lymphocytes (TIL) clone DMF5.

We constructed a single retroviral vector that encodes both alpha and beta chains and can mediate genetic transfer of this T cell receptor (TCR) with high efficiency without the need to perform any selection.

In co-cultures with HLA-A*0201 positive melanoma, anti-MART-1 F5 TCR transduced T cells secreted significant amount of IFN- but no significant secretion was observed in control co-cultures with cell lines.

The anti-MART-1 F5 TCR transduced PBL could efficiently kill HLA-A*0201 positive tumors. There was little or no recognition of normal fibroblasts cells.

This TCR is over 10 times more reactive with melanoma cells than the MART-1 F4 TCR that mediated tumor regression in two patients with metastatic melanoma.

Poxviruses encoding melanoma antigens, similar to the ALVAC MART-1 vaccine have been shown to successfully immunize patients against these antigens.

Objectives:

Primary objectives:

To evaluate the ability of four different strategies to enhance the persistence of anti-tumor T cells in the circulation at 5-10 days, and at 31-35 days after treatment (defined as F5 cells in cohorts 1 and 2, and aldesleukin in cohorts 3 and 4) and potentially select one strategy for further study.

With Amendment E, the primary objective is to evaluate the ability of three different strategies to enhance the persistence of anti-tumor T cells in the circulation at 5-10 days and at 31-35 days after treatment (defined as F5 cells in cohort 5, aldesleukin in cohort 6, and ALVAC MART-1 vaccine in cohort 7) and potentially select one strategy for further study.

Eligibility:

Patients who are HLA-A*0201 positive and 18 years of age or older must have:

* primary melanomas with lesions that are ulcerated and greater than or equal to 2.0 mm, or any lesions that are greater than or equal to 4.0 mm in thickness, or greater than or equal to 1 positive lymph node, or local recurrence, or resected metastatic disease, within 6 months of surgical resection.
* must be clinically disease free at the time of protocol entry as documented by radiologic studies within 4 weeks of patient entry.
* may have had prior adjuvant treatment with immunotherapy, including interferon, as long as 3 weeks have elapsed since prior systemic therapy.
* normal values for basic laboratory values.

Patients may not have:

* ocular or mucosal melanoma;
* been previously immunized with MART-1;
* concurrent major medical illnesses;
* any form of primary or secondary immunodeficiency;
* severe hypersensitivity to any of the agents used in this study;

Design:

Peripheral blood mononuclear cells (PBMC) obtained by leukapheresis (approximately 1 times 10^10 cells) will be cultured in the presence of anti-CD3 (OKT3) and aldesleukin in order to stimulate T-cell growth.

Transduction is initiated by exposure of approximately 10^8 to 5 times 10^9 cells to retroviral vector supernatant containing the anti-MART-1 F5 TCR genes. These transduced cells (called F5 cells) will be expanded and tested for their anti-tumor activity.

F5 cells will be administered intravenously at a dose of 1 times 10^9 to 7 times 10^10 cells.

Patients will be randomized into one of the following four cohorts:

1. F5 cells on day 0 alone
2. F5 cells on day 0 followed by the subcutaneous injection of 1.0 mg MART-1:26-35(27L) peptide in Montanide ISA-51 VG on day 0 and day 30.
3. F5 cells on day 0 followed by the subcutaneous injection of 125,000 IU/kg/day aldesleukin on days 0-4.
4. F5 cells on day 0 plus MART-1:26-35(27L) peptide in Montanide ISA-51 VG on day 0 and day 30, and 125,000 IU/kg aldesleukin on days 0-4.

   Starting with amendment E, the four cohorts above will be closed to accrual and patients will be randomized to the following cohorts:
5. F5 cells on day 0 following subcutaneous injection of ALVAC MART-1 vaccine. Second dose of ALVAC MART-1 vaccine is given on day 14.
6. F5 cells on day 0 following subcutaneous injection of ALVAC MART-1 vaccine and then subcutaneous injection of 125,000 IU/kg/day aldesleukin on days 0-4. Second dose of ALVAC MART-1 vaccine is given on day 14.
7. ALVAC MART-1 vaccine on days 0 and 14.

Patients will undergo complete evaluation with physical examination, computed tomography (CT) of the chest, abdomen and pelvis (3 months and thereafter only) and clinical laboratory evaluation at day 35, and 3 months after treatment and then every six months or until off study criteria are met.

Each of the cohorts will be conducted using a two-stage MiniMax design. This design will try to determine whether each of the modalities of administration can produce persistence of the transferred cells at a frequency of greater than or equal to 5 percent of circulating cluster of differentiation 8 (CD8) plus cells in 35 percent of patients as opposed to undesirably low (15 percent), with a 3 percent probability of accepting a poor schedule and 15 percent probability of rejecting a good schedule.

Initially 22 patients will be enrolled in each cohort. If four immunologic responses (persistence) are noted in a given cohort, then accrual to 39 patients would take place. The cohort with the highest number of patients exhibiting persistence will be considered immunologically active and will be considered worthy of further development. If this arm has fewer than 11 of 39 patients with persistence, it will not be considered worthy of further consideration.

Starting with amendment E, 10 patients will be enrolled in each new cohort (cohorts 5-7). If on any of the three arms, there are 2 or more of 10 patients with 5% CD8+ circulating cells, then this cohort will be considered worthy of further consideration.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Primary melanomas with lesions that are ulcerated and greater than or equal to 2.0 mm, or any lesions that are greater than or equal to 4.0 mm in thickness, or greater than or equal to 1 positive lymph node, or local recurrence, or resected metastatic disease, within 6 months of surgical resection will be considered. Patients must be clinically disease free at the time of protocol entry as documented by radiologic studies within 6 weeks of patient entry. Patients must have pathologic confirmation of cutaneous melanoma, with slides reviewed at National Institutes of Health (NIH) (Department of Anatomic Pathology), and if the diagnosis is not confirmed, the patient will be excluded from the study.
  2. Human leukocyte antigens (HLA-A) 0201 positive.
  3. Age greater than or equal to18 years.
  4. Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0 or 1.
  5. Able to understand and sign the Informed Consent Document.
  6. Patients of both genders must be willing to practice effective birth control during this trial because the potential for teratogenic effects are unknown. Effective birth control requires use of an effective method from the following list: Abstinence, Intrauterine device (IUD); Hormonal (Birth control pills, injections, implants); Tubal ligation; Cervical cap; or Partner's vasectomy
  7. Patients may have had prior adjuvant treatment with immunotherapy, including interferon, as long as 3 weeks have elapsed since prior systemic therapy.
  8. Serology:

     1. Seronegative for human immunodeficiency virus (HIV) antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune -competence and thus be less responsive to the experimental treatment and more susceptible to its toxicities.)
     2. Seronegative for hepatitis B antigen and hepatitis C antibody unless antigen negative (The experimental treatment being evaluated in this protocol depends upon an intact immune system and these conditions may have possible immune system effects).
  9. Hematology:

     1. Absolute neutrophil count greater than 1000/mm^3 without the support of filgrastim.
     2. White blood cell (WBC) (greater than 3000/mm^3).
     3. Platelet count greater than 90,000/mm^3.
     4. Hemoglobin greater than 8.0 g/dl.
  10. Chemistry:

      1. Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) less or equal to 2.5 times the upper limit of normal.
      2. Serum creatinine less than or equal to 1.6 mg/dl.
      3. Total bilirubin less than or equal to 1.5 mg/dl, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dl.

EXCLUSION CRITERIA:

1. Ocular or mucosal melanoma.
2. Undergoing or have undergone in the past 3 weeks any systemic therapy except surgery for their cancer, and must have recovered to a grade 1 from any adverse effects of treatment prior to entry, other than those that do not have clinical implications, e.g. vitiligo, alopecia.
3. Have autoimmune disease (such as autoimmune colitis or Crohn's disease) or any known immunodeficiency disease, as evidenced by abnormal white blood count (WBC) count.
4. Concurrent systemic steroid therapy.
5. Known systemic hypersensitivity to any of the vaccine components, including egg products or Neomycin.
6. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the treatment on the fetus or infant.
7. Have active systemic infections including concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities).
8. Previous immunization with melanoma antigen recognized by T cells (MART-1).
9. Known hypersensitivity to any of the agents used in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-06; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Rosenberg, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Schwartz RH. T cell clonal anergy. Curr Opin Immunol. 1997 Jun;9(3):351-7. doi: 10.1016/s0952-7915(97)80081-7. PMID 9203408
- [Background] Rosenberg SA, Yang JC, Restifo NP. Cancer immunotherapy: moving beyond current vaccines. Nat Med. 2004 Sep;10(9):909-15. doi: 10.1038/nm1100. PMID 15340416
- [Background] Dudley ME, Wunderlich JR, Robbins PF, Yang JC, Hwu P, Schwartzentruber DJ, Topalian SL, Sherry R, Restifo NP, Hubicki AM, Robinson MR, Raffeld M, Duray P, Seipp CA, Rogers-Freezer L, Morton KE, Mavroukakis SA, White DE, Rosenberg SA. Cancer regression and autoimmunity in patients after clonal repopulation with antitumor lymphocytes. Science. 2002 Oct 25;298(5594):850-4. doi: 10.1126/science.1076514. Epub 2002 Sep 19. PMID 12242449

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm III - Adj-4 A2 F5 Cells + SQ IL-2: Patients receive anti-MART-1 F5 TCR-transduced PBLs as in arm I and aldesleukin SC on days 0-4. 1 x 10e9 to 5 x 10e10 IV + IL-2 (based on body weight) 125,000 IU/kg/day subcutaneously.
- Arm IV-Adj-4 A2 F5 Cells + MART-1:26-35(27L) Peptide + SQ IL-2: Patients receive anti-MART-1 F5 TCR-transduced PBLs as in arm I, MART-1:26-35(27L) peptide vaccine emulsified in Montanide ISA-51 as in arm II, and aldesleukin as in arm III. 1 x 10e9 to 5 x 10e10 IV + 1.0 mg peptide subcutaneously + IL-2 (based on body weight) 125,000 IU/kg/day subcutaneously.
- Arm VII - Adj-4 A2 ALVAC MART-1 Vaccine: Patients receive ALVAC-MART-1 vaccine SC on days 0 and 14. ALVAC vaccine 0.5 ml containing target dose of 10e7 CCID50 (with a range of approximately 10^6.4 to 10^7.9/mL subcutaneously (total of 4 x 10e7 CCID50/2 mL).
Period: Overall Study
Arm/Group | Arm I - Adj-4 A2 F5 Cells | Arm II-Adj-4 A2 F5 Cells + MART-1:26-35(27L) Peptide | Arm III - Adj-4 A2 F5 Cells + SQ IL-2 | Arm IV-Adj-4 A2 F5 Cells + MART-1:26-35(27L) Peptide + SQ IL-2 | Arm V-Adj-4 A2 F5 Cells + ALVAC MART-1:26-35(27L) Vaccine | Arm VI-Adj-4 A2 F5 Cells + ALVAC MART-1 Vaccine + SQ IL-2 | Arm VII - Adj-4 A2 ALVAC MART-1 Vaccine
Started | 8 | 8 | 9 | 8 | 6 | 5 | 6
Completed | 3 | 3 | 3 | 6 | 2 | 3 | 3
Not Completed | 5 | 5 | 6 | 2 | 4 | 2 | 3
Not completed — Study termination | 5 | 5 | 6 | 2 | 3 | 2 | 3
Not completed — Disease progression before treatment | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm I: Patients receive anti-MART-1 F5 TCR-transduced peripheral blood lymphocytes (PBLs) intravenously (IV) over 20-30 minutes on day 0. 1 x 10e9 to 5 x 10e10 IV.
- Arm II: Patients receive anti-MART-1 F5 TCR-transduced PBLs as in arm I and MART-1:26-35(27L) peptide vaccine emulsified in Montanide ISA-51 subcutaneously (SC) on days 0 and 30. 1 x 10e9 to 5 x 10e10 IV + 1.0 mg peptide subcutaneously.
- Arm III: Patients receive anti-MART-1 F5 TCR-transduced PBLs as in arm I and aldesleukin SC on days 0-4. 1 x 10e9 to 5 x 10e10 IV + IL-2 (based on body weight) 125,000 IU/kg/day subcutaneously.
- Arm IV: Patients receive anti-MART-1 F5 TCR-transduced PBLs as in arm I, MART-1:26-35(27L) peptide vaccine emulsified in Montanide ISA-51 as in arm II, and aldesleukin as in arm III. 1 x 10e9 to 5 x 10e10 IV + 1.0 mg peptide subcutaneously + IL-2 (based on body weight) 125,000 IU/kg/day subcutaneously.
- Arm V: Patients receive anti-MART-1 F5 TCR-transduced PBLs IV over 20-30 minutes on day 0, and ALVAC-MART-1 vaccine SC on days 0 and 14. 1 x 10e9 to 5 x 10e10 IV + ALVAC vaccine 0.5 ml containing target dose of 10e7 CCID50 (with a range of approximately 10^6.4 to 10^7.9/mL subcutaneously (total of 4 x 10e7 CCID50/2 mL).
- Arm VI: Patients receive anti-MART-1 F5 TCR-transduced PBLs and ALVAC-MART-1 vaccine as in arm V, and low-dose aldesleukin SC on days 0-4. 1 x 10e9 to 5 x 10e10 IV + ALVAC vaccine 0.5 ml containing target dose of 10e7 CCID50 (with a range of approximately 10^6.4 to 10^7.9/mL subcutaneously (total of 4 x 10e7 CCID50/2 mL)+ 125,000 IU/kg/day subcutaneously.
- Arm VII: Patients receive ALVAC-MART-1 vaccine SC on days 0 and 14. ALVAC vaccine 0.5 ml containing target dose of 10e7 CCID50 (with a range of approximately 10^6.4 to 10^7.9/mL subcutaneously (total of 4 x 10e7 CCID50/2 mL).
- Total: Total of all reporting groups
Arm/Group | Arm I | Arm II | Arm III | Arm IV | Arm V | Arm VI | Arm VII | Total
Number analyzed (Participants) | 8 | 8 | 9 | 8 | 6 | 5 | 6 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 9 | 8 | 6 | 5 | 6 | 50
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.0 (12.9) | 47.4 (8.9) | 43.1 (11.4) | 51.4 (9.7) | 49.2 (8.3) | 49.0 (11.2) | 39.2 (5.7) | 47.2 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 5 | 1 | 3 | 1 | 3 | 20
  Male | 4 | 5 | 4 | 7 | 3 | 4 | 3 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 8 | 7 | 9 | 8 | 6 | 5 | 6 | 49
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  White | 8 | 7 | 8 | 8 | 6 | 5 | 6 | 48
  More than one race | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 9 | 8 | 6 | 5 | 6 | 50

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Immunologic Response
Description: Percentage of participants with an immunologic response of >20 spots/100,000 cells measured by IFN gamma secretion using enzyme linked immunosorbent spot (ELISPOT) assay. This was done using ELISPOT assay which measures immune response at the single cell level.
Time Frame: 9/24/08-10/9/12
Population: Arms 1-6 were evaluated in patients who received F5 cells. Arm 7 was not included in the evaluation because the participants did not receive F5 cells.The immunological response was measured for the total percentage of pts whom specimen was available for analysis. This was not captured per Arm. No statistically significant responses were observed.
Measure: Number; unit: Percentage of participants
Groups:
- Arm I - 6: Arm I - Adj-4 A2 F5 cells Arm II-Adj-4 A2 F5 cells + MART-1:26-35(27L) Peptide Arm III-Adj-4 A2 F5 cells + SQ IL-2 Arm IV-Adj-4 A2 F5 cells + MART-1:26-35(27L) Peptide+SQ IL-2 Arm V-Adj-4 A2 F5 cells + ALVAC MART-1:26-35(27L) Vaccine Arm VI-Adj-4 A2 F5 cells + ALVAC MART-1 Vaccine + SQ IL-2
Arm/Group | Arm I - 6
Number analyzed (Participants) | 40
Percentage of participants | 0

2. Primary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For a detailed list of adverse events see the adverse event module.
Time Frame: 4 years
Measure: Number; unit: Participants
Arm/Group | Arm I - Adj-4 A2 F5 Cells | Arm II-Adj-4 A2 F5 Cells + MART-1:26-35(27L) Peptide | Arm III - Adj-4 A2 F5 Cells + SQ IL-2 | Arm IV-Adj-4 A2 F5 Cells + MART-1:26-35(27L) Peptide + SQ IL-2 | Arm V-Adj-4 A2 F5 Cells + ALVAC MART-1:26-35(27L) Vaccine | Arm VI-Adj-4 A2 F5 Cells + ALVAC MART-1 Vaccine + SQ IL-2 | Arm VII - Adj-4 A2 ALVAC MART-1 Vaccine
Number analyzed (Participants) | 8 | 8 | 9 | 8 | 6 | 5 | 6
Participants | 8 | 7 | 8 | 8 | 4 | 5 | 1

ADVERSE EVENTS:
Arm/Group | Arm I | Arm II | Arm III | Arm IV | Arm V | Arm VI | Arm VII
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/9 | 0/8 | 0/6 | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 8/8 | 7/8 | 8/9 | 8/8 | 4/6 | 5/5 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=8) | Arm II (N=8) | Arm III (N=9) | Arm IV (N=8) | Arm V (N=6) | Arm VI (N=5) | Arm VII (N=6)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 7 (7) | 1 (1) | 7 (7) | 5 (5) | 4 (4) | 3 (3) | 0 (0)
Urticaria (hives, welts, wheals) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OCULAR/VISUAL:: Ocular/Visual-Other, left conjunctivitis (inflammation) (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain - Other, body aches (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 5 (5) | 7 (7) | 0 (0) | 5 (5) | 0 (0)
Rigors/chills (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Injection site reaction/extravasation changes (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (6) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Pain (General disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (4) | 0 (0) | 1 (1) | 0 (0)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutropenia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 3 (3) | 0 (0)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 5 (5) | 0 (0) | 3 (3) | 0 (0)
Psychosis (hallucinations/delusions) (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision-blurred vision (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
OCULAR/VISUAL:: Ocular/Visual-Other (Specify) (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Decreased vision; Blurry vision due to retinal edema
Pain - Other, body pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal - Other, sigmoid diverticulosis (incidental finding on CT scan) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alkaline phosphatase (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OCULAR/VISUAL:: Ocular/Visual-Other, vision changes (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uveitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Creatinine (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No